CLINICAL TRIAL: NCT04770441
Title: Prospective Evaluation of the Use of TIF (Transoral Incisionless Fundoplication) to Treat Post-poem GERD
Brief Title: Transoral Incisionless Fundoplication in Post-POEM GERD
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Salmaan Azam Jawaid, MD, Principal Investigator, Baylor College of Medicine
Other Study IDs: H-48496
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Swallowing Disorders; Achalasia; Outlet Obstruction, Gastric; Diffuse Esophageal Spasm
Keywords: Per-Oral Endoscopic Myotomy (POEM); Submucosal Endoscopy
MeSH Terms: conditions — Deglutition Disorders; Esophageal Achalasia; Gastric Outlet Obstruction; Esophageal Spasm, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
POEM (per oral endoscopic myotomy) is effective for the treatment of swallowing disorders but can induce acid reflux. If acid reflux remains untreated in this situation, it can lead to significant problems. Thus, minimizing abnormal acid exposure after POEM is very important. Typically, this is done with acid suppression medications such as Prilosec or Nexium. However, long term acid suppression medication has been linked to possible long-term complications. Transoral incisionless fundoplication (TIF) has been approved for the treatment of reflux, but its use in reflux after POEM has not been investigated in detail. We hypothesize TIF will be able to decrease the amount of acid reflux in to the esophagus, thereby allowing patients to remain off of acid suppression medications.

Once enrolled into the study, you will undergo the POEM procedure. 3 months after the procedure we will assess for abnormal reflux via questionnaires and diagnostic testing as part of the standard management post POEM. If there is evidence of abnormal reflux, the TIF procedure will be performed. 3 months after the TIF, you will have similar testing again to document resolution in abnormal acid reflux.You will be followed for 12 months as part of the study. If at the 3 month mark, there is no evidence of abnormal reflux, you will neither be placed on PPI nor undergo TIF and will be followed for 12 months to assess for abnormal reflux

DETAILED DESCRIPTION:
EGD (esophagogastroduodenoscopy) is a safe procedure used extensively to evaluate the esophagus, stomach and small intestine. With the assistance of the anesthesiology team, we will put you to sleep partially to minimize discomfort during the insertion of the endoscopy. This is normally how this procedure is performed and deemed very safe. Potential complications include breathing problems, holes in the intestine, and bleeding. These occur very infrequently. In our study, EGD will be used at three checkpoints (all of which are part of standard of care):

1. at the time of POEM to rule out other unusual structural abnormalities
2. at 3 months during measurement of acid exposure in the esophagus via Bravo pH
3. 3 months after TIF placement (6 months after enrollment and POEM) to document resolution in acid reflux.

Esophageal manometry is a non-endoscopic procedure that involves using a safe numbing cream to allow passage of the manometry catheter from the nose down to the end of the esophagus. Different measurements are taken from the catheter and the catheter is then removed. This is a standard of care procedure in the evaluation of patients with esophageal motility/swallowing disorders. It will be used in the following settings and all are part of standard of care:

1. 3 months after POEM as part of standard of care to assess improvement in the swallowing
2. 3 months after TIF (6 months post POEM) only if swallowing issues reappear.

Bravo pH study is used to assess abnormal acid reflux and is considered gold standard in identifying the degree of acid reflux. It is standard of care for this procedure to be performed in patients with suspected acid reflux and post-POEM to assess need for long term acid suppression. It involves performing an endoscopy first, followed by deployment and implantation of the Bravo pH capsule into the end of the esophagus. Risks include bleeding, injury to the esophagus or dislodgment of the capsule. However, these are rare instances.

POEM Those enrolled into the study will undergo a diagnostic endoscopy at the same allotted time as the POEM. It will be explained to you in detail but involves endoscopically cutting the muscle at the end of the esophagus, called a myotomy. It is less invasive than its surgical equivalent Heller's myotomy, but equally effective. Two endoscopist (one with extensive experience in POEM and the other with formal training in POEM) will be performing the actual POEM procedures.

TIF The TIF procedure is performed using the FDA approved EsophyX-Z device (EndoGastricSolutions, Redmond, Wash, USA). It has been shown to be effective in the management of acid reflux in patients who fail acid suppression therapy or in patients who would like to avoid long term acid suppression with acid suppression therapy due to the potential side effects. It involves the use of a flexible suturing apparatus that fits over the endoscope and is used to create an artificial wrap around the end of the esophagus, thereby mimicking the effects of the typical surgical wrap. In the right setting it is as effective as its surgical counterpart but less invasive. Due to the incisionless approach, patients undergoing TIF experience less discomfort and faster recovery than those undergoing traditional anti-reflux surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years old
* Able to sign consent
* Patients must meet standard clinical indications for POEM procedure (all indications) for the initial enrollment
* To undergo TIF: Evidence of GERD/GERD related complications after POEM:
* pathologic acid exposure on pH testing (Deemester score >14.72 or percentage time pH <4 greater than 5.3%) off of PPI (19)
* esophagitis on EGD (grades A to C)
* biopsies showing evidence of reflux esophagitis

Exclusion Criteria:

* Adults unable to consent
* Pregnant women - Prisoners
* Delayed gastric emptying
* Code status of DNR/DNI or CMO
* Any patient with moderate to severe esophagitis pre-POEM
* Grade D esophagitis post POEM
* Hiatal hernia >2cm
* PPI use prior to POEM (and if PPI is needed)
* Previous surgery of the stomach
* Known GI malignancy
* Cirrhosis with portal hypertension, varices, or ascites
* Previous anti-reflux surgery
* Patients who choose not to undergo TIF or if insurance will not cover the procedure.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with confirmed indications for POEM (achalasia, jackhammer esophagus, EGJOO, diffuse esophageal spasm) will be identified as potential study patients. These patients will undergo objective testing and will be required to complete subjective questionnaires for achalasia and GERD as part of the standard work up (off of PPI therapy). Additionally, chart review of their medical records will be conducted for clinical outcomes. These include: - pre-POEM esophageal manometry and pH testing - GERD-HRQL (separate heartburn and regurgitation scores) - Eckardt scores - EGD pre-POEM (patients will be assessed for hiatal hernia as documented by length, diameter, and Hill grade)
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2023-06-03 (Actual)

PRIMARY OUTCOMES:
Percentage of patients not requiring PPI therapy at set endpoints | 1 year
  If at least 50% of patients do not require initiation of PPI therapy at the end of the study, then TIF would be considered successful.

SECONDARY OUTCOMES:
At least 50% of patients with a 50% decrease in GERD-HQRL 3 months post TIF (20) | 1 year
  Assessed and evaluated at protocol's scheduled visits.
Decrease in Demeester scores to less than 14.72 (above this number is consider pathologic acid reflux) in at least 50% of patients | 1 year
  Assessed and evaluated at protocol's scheduled visits.
50% decrease in the number of patients with percentage of time of acid exposure (pH <4) was less than or equal to 5.3% | 1 year
  Assessed and evaluated at protocol's scheduled visits.
50% decrease in the number of patients with percentage time pH <4 reduced to 30% of the pre-TIF value (21) | 1 year
  Assessed and evaluated at protocol's scheduled visits.
50% improvement in esophageal GERD related | 1 year
  Assessed and evaluated at protocol's scheduled visits.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
This is a single-site prospective study.